CLINICAL TRIAL: NCT07158047
Title: Targeting Hypertension and Insulin Resistance With Heat Therapy
Brief Title: Repeated Far Infrared Sauna Bathing in Adults With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Christopher T Minson, PhD, Professor, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07312020.034; 19TPA34890033 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obesity (Disorder)
Keywords: heat therapy; insulin resistance; arterial stiffness; blood pressure; obesity; sauna; vascular health; cardiovascular; metabolic function
MeSH Terms: conditions — Obesity; Hyperthermia; Insulin Resistance | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Time control versus heat therapy group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat therapy (Experimental): Group will undergo 30 sessions of heat therapy over approximately 10 weeks. Sessions will require participants to sit in a far infrared sauna for up to 45 min for 3 to 4 times per week.
  Interventions: Other: Heat therapy
- Time control group (No Intervention): No participation in sauna bathing. Maintain lifestyle habits for approximately 10 weeks.

INTERVENTIONS:
Other: Heat therapy — 30 sessions of far infrared sauna bathing (45-60C) for up to 45 min
  Other Names: sauna bathing
  Arms: Heat therapy

SUMMARY:
This is a clinical trial to determine if 30 sessions of far infrared sauna bathing can improve cardiovascular and metabolic function in adults with obesity.

DETAILED DESCRIPTION:
Obesity can increase the risk for cardiovascular and metabolic diseases. Lifestyle interventions are needed to reduce this risk. Far infrared saunas are one form of heat therapy that may help reduce these risks, however, there is limited research within a population with obesity. It is hypothesized that repeated far infrared sauna bathing will improve cardiovascular and metabolic function in adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-45 kg/m2

Exclusion Criteria:

* Diagnosed diabetes
* Greater than stage 2 hypertension
* Coagulopathies
* Allergies to lidocaine
* Medications affecting blood pressure
* Blood clotting, and blood sugars
* Smoker
* Pregnant
* Desiring to become pregnant in the near future
* Breastfeeding
* BMI less than 30
* BMI greater than 45 kg/m2
* Exercising > 120 min/week
* Taking medications (other than hormone contraceptives)
* Not willing to stop taking medications (other than hormone contraceptives) for 24 hours before testing days

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change | 10 weeks
  Change in systolic and diastolic blood pressures after 30 sessions of Intervention
Blood glucose | 10 weeks
  Change in plasma glucose levels after Intervention

SECONDARY OUTCOMES:
Arterial stiffness reduction | 10 weeks
  Change in Carotid-femoral Pulse Wave Velocity (m/s) after Intervention
Serum insulin | 10 weeks
  Change in serum insulin levels after Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Minson, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masuda A, Koga Y, Hattanmaru M, Minagoe S, Tei C. The effects of repeated thermal therapy for patients with chronic pain. Psychother Psychosom. 2005;74(5):288-94. doi: 10.1159/000086319. PMID 16088266
- [Background] Kihara T, Biro S, Imamura M, Yoshifuku S, Takasaki K, Ikeda Y, Otuji Y, Minagoe S, Toyama Y, Tei C. Repeated sauna treatment improves vascular endothelial and cardiac function in patients with chronic heart failure. J Am Coll Cardiol. 2002 Mar 6;39(5):754-9. doi: 10.1016/s0735-1097(01)01824-1. PMID 11869837
- [Background] Kihara T, Biro S, Ikeda Y, Fukudome T, Shinsato T, Masuda A, Miyata M, Hamasaki S, Otsuji Y, Minagoe S, Akiba S, Tei C. Effects of repeated sauna treatment on ventricular arrhythmias in patients with chronic heart failure. Circ J. 2004 Dec;68(12):1146-51. doi: 10.1253/circj.68.1146. PMID 15564698
- [Background] Fuchs CJ, Betz MW, Petrick HL, Weber J, Senden JM, Hendriks FK, Bels JLM, van Loon LJC, Snijders T. Repeated passive heat treatment increases muscle tissue capillarization, but does not affect postprandial muscle protein synthesis rates in healthy older adults. J Physiol. 2025 Jan;603(1):167-186. doi: 10.1113/JP286986. Epub 2024 Oct 7. PMID 39373667
- [Background] Ely BR, Francisco MA, Halliwill JR, Bryan SD, Comrada LN, Larson EA, Brunt VE, Minson CT. Heat therapy reduces sympathetic activity and improves cardiovascular risk profile in women who are obese with polycystic ovary syndrome. Am J Physiol Regul Integr Comp Physiol. 2019 Nov 1;317(5):R630-R640. doi: 10.1152/ajpregu.00078.2019. Epub 2019 Sep 4. PMID 31483156
- [Background] Ely BR, Clayton ZS, McCurdy CE, Pfeiffer J, Needham KW, Comrada LN, Minson CT. Heat therapy improves glucose tolerance and adipose tissue insulin signaling in polycystic ovary syndrome. Am J Physiol Endocrinol Metab. 2019 Jul 1;317(1):E172-E182. doi: 10.1152/ajpendo.00549.2018. Epub 2019 May 28. PMID 31136202
- [Background] Brunt VE, Jeckell AT, Ely BR, Howard MJ, Thijssen DH, Minson CT. Acute hot water immersion is protective against impaired vascular function following forearm ischemia-reperfusion in young healthy humans. Am J Physiol Regul Integr Comp Physiol. 2016 Dec 1;311(6):R1060-R1067. doi: 10.1152/ajpregu.00301.2016. Epub 2016 Oct 5. PMID 27707723
- [Background] Brunt VE, Eymann TM, Francisco MA, Howard MJ, Minson CT. Passive heat therapy improves cutaneous microvascular function in sedentary humans via improved nitric oxide-dependent dilation. J Appl Physiol (1985). 2016 Sep 1;121(3):716-23. doi: 10.1152/japplphysiol.00424.2016. Epub 2016 Jul 14. PMID 27418688
- [Background] Behzadi P, Ravanelli N, Gravel H, Barry H, Debray A, Chaseling GK, Jacquemet V, Neagoe PE, Nigam A, Carpentier AC, Sirois MG, Gagnon D. Acute effect of passive heat exposure on markers of cardiometabolic function in adults with type 2 diabetes mellitus. J Appl Physiol (1985). 2022 May 1;132(5):1154-1166. doi: 10.1152/japplphysiol.00800.2021. Epub 2022 Mar 24. PMID 35323077